CLINICAL TRIAL: NCT01950104
Title: Comparative Study Between Day 3 Embryo Biopsy and Blastocyst Biopsy in Preimplantation Genetic Screening Cases
Brief Title: Day 3 Embryo Biopsy Versus Blastocyst Biopsy in PGS Cases
Acronym: VINCI
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No started, lack of funding
Sponsor: Vida Recoletas Sevilla (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IVISEV-005VINCI
Record Dates: First submitted 2013-09-23; First posted 2013-09-25 (Estimated); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Infertility; Embryo Biopsy
Keywords: Embryo biopsy; Blastocyst stage; Day 3; Preimplantation genetic screening
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Day 3 embryo biopsy (Active Comparator): Embryo biopsy is applied at day 3 of the embryo development
  Interventions: Other: Day 3 embryo biopsy
- Blastocyst biopsy (Experimental): Embryo biopsy is applied at the blastocyst stage of the embryo development (day 5 or 6)
  Interventions: Other: Blastocyst biopsy

INTERVENTIONS:
Other: Day 3 embryo biopsy — Embryo biopsy is applied at day 3 of the embryo development.
  Arms: Day 3 embryo biopsy
Other: Blastocyst biopsy — Embryo biopsy is applied at the blastocyst stage of the embryo development
  Arms: Blastocyst biopsy

SUMMARY:
Preimplantation genetic diagnosis (PGS) is a technique that allow us to improve the results of assisted reproduction techniques through the selection of embryos free of chromosomal abnormalities.

At present, it has not been proved that the usage of PGS really improves the live birth rate in IVF cycles. However, it has been stated that the reason of not having better results when using PGS is that the methodology applied is not adequate.

Several authors propose that the optimal methodology for PGS includes the application of comparative genomic hybridization (CGH) arrays for genetic testing and carrying out embryo biopsy at the blastocyst stage. Nevertheless, most IVF centres still applies the day 3 embryo biopsy as a daily routine. Despite this fact, there is a gradual transition towards the usage of blastocyst-stage biopsy instead of day 3 biopsy.

The purpose of this clinical study is analysing the results of the IVF cycles with embryo biopsy for PGS. Live birth rates and other parameters as the pregnancy and implantation rates together with embryo quality will be analysed and compared between two groups of patients undergoing IVF cycles with PGS. In one group the biopsy will be applied in day 3 of the embryo development, while in the other group the embryo biopsy will be fulfilled at the blastocyst stage.

ELIGIBILITY:
Inclusion Criteria:

Patients under 49 years undergoing IVF cycles with PGS for one of the following reasons:

* Advanced maternal age
* Recurrent implantation failure
* Recurrent abortion
* Severe male-factor infertility

Exclusion Criteria:

* Not being able to sign the informed consent to participate in the study
* Patients undergoing preimplantation genetic diagnosis

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Live birth rate | 20 months

SECONDARY OUTCOMES:
Fertilization rate | 1 year
Embryo quality | 1 year
  Day 3 embryo quality
Implantation rate | 1 year
Pregnancy rate | 20 months

CONTACTS AND LOCATIONS:
Locations (1):
- IVI Sevilla, Seville, Spain